CLINICAL TRIAL: NCT04738708
Title: Telegenetics or In-Person Genetic Counselling: A Comparison of Clinical Outcomes and Cost
Brief Title: Telegenetics or In-Person Genetic Counselling
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 002.1
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Genetic Counselling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred to CGS at NCCS for HBOC or Lynch syndrome pre-test genetic counselling.: Patients attending genetic counselling for Hereditary Breast and Ovarian Cancer (HBOC) and Lynch Syndrome in Clinical Genetic Services (CGS) at National Cancer Centre Singapore (NCCS)
  Interventions: Other: Patients referred to CGS at NCCS for HBOC or Lynch syndrome pre-test genetic counselling.

INTERVENTIONS:
Other: Patients referred to CGS at NCCS for HBOC or Lynch syndrome pre-test genetic counselling. — Patients are given a series of questions evaluating cognitive and psychosocial outcomes, either via hardcopy in-person or online internet-facing questionnaire.

SUMMARY:
This study aims to compare clinical outcomes (informed choice and genetic counselling outcomes) and cost (provider and patient time, travel, and telehealth platform) between telegenetics and in-person genetic counselling.

DETAILED DESCRIPTION:
This study will compare the patient-reported outcomes of telegenetics with in-person consultations for participants considering germline testing for HBOC or Lynch syndrome. It will clarify if telegenetics is a feasible and non-inferior alternative to in-person cancer genetic counselling. Participant responses are important stakeholder views to guide the design of telegenetics to become a mainstream service delivery model welcomed by patients.

It aims to recruit 150 prospective consecutive patients attending genetic counselling for Hereditary Breast and Ovarian Cancer (HBOC) and Lynch Syndrome in Clinical Genetic Services (CGS) at National Cancer Centre Singapore (NCCS).

Upon completion of the genetic consultation appointments, patients will be completing a series of questions evaluating cognitive and psychosocial outcomes either via hardcopy in-person or online internet-facing questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years old.
* Patients referred to CGS at NCCS for HBOC or Lynch syndrome pre-test genetic counselling.
* Able to read and understand the English Language.
* Able to consent and agree to be randomized to either telegenetics or in-person genetic counselling.

Exclusion Criteria:

* Under the age of 21 years old.
* Patients who require genetic results urgently.
* Cognitive difficulty/ impairment or current psychiatric or physical illness (visual/ hearing/ neurological) which impairs sound judgement and accurate reporting of medical history over video consultation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to CGS at NCCS for HBOC or Lynch syndrome pre-test genetic counselling.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Genomics Outcome Scale | Up to 2 weeks after consultation
  Patient reported outcomes will be compared with a 6 item Genomics Outcome Scale (GOS) across five domains (decisional control, cognitive control, behavioral control, emotional regulation and hope) which are rated on a 5-point Likert scale ranging from "strongly agree" to "strongly disagree". Scores are summed to provide an overall "empowerment" where higher scores equal higher levels of empowerment.

SECONDARY OUTCOMES:
Adapted Multidimensional Measure of Informed Choice (MMIC) for Hereditary Breast and Ovarian Cancer (HBOC) and Lynch | Up to 2 weeks after consultation
  Participant's knowledge and attitude of HBOC and Lynch syndrome will be compared with a multi-dimensional measure of informed choice (MMIC) which composed of 11 items for knowledge of HBOC or 12 items for knowledge of Lynch syndrome and 4 items for attitudes. Items will be summed with a score or rated on a 7-pointed Likert scale.
Genetic Counselling Satisfaction Scale | Up to 2 weeks after consultation
  Genetic counselling satisfaction is measured with a 6 item Genetic Counselling Satisfaction Scale. Items will be rated on a 5-point Likert scale and summed. Higher scores indicating higher satisfaction.
Telehealth Patient Survey | Up to 2 weeks after consultation
  Telehealth satisfaction is measured with a 7 item Telehealth Patient Survey. Items will be rated on a 5-point Likert scale and summed. Higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Tan, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

REFERENCES:
- [Background] Lee AKF, Cho RHW, Lau EHL, Cheng HK, Wong EWY, Ku PKM, Chan JYK, Yeung ZWC. Mitigation of head and neck cancer service disruption during COVID-19 in Hong Kong through telehealth and multi-institutional collaboration. Head Neck. 2020 Jul;42(7):1454-1459. doi: 10.1002/hed.26226. Epub 2020 May 7. PMID 32357277
- [Background] Lonergan PE, Washington Iii SL, Branagan L, Gleason N, Pruthi RS, Carroll PR, Odisho AY. Rapid Utilization of Telehealth in a Comprehensive Cancer Center as a Response to COVID-19: Cross-Sectional Analysis. J Med Internet Res. 2020 Jul 6;22(7):e19322. doi: 10.2196/19322. PMID 32568721
- [Background] Pramesh CS, Badwe RA. Cancer Management in India during Covid-19. N Engl J Med. 2020 May 14;382(20):e61. doi: 10.1056/NEJMc2011595. Epub 2020 Apr 28. No abstract available. PMID 32343498
- [Background] van de Haar J, Hoes LR, Coles CE, Seamon K, Frohling S, Jager D, Valenza F, de Braud F, De Petris L, Bergh J, Ernberg I, Besse B, Barlesi F, Garralda E, Piris-Gimenez A, Baumann M, Apolone G, Soria JC, Tabernero J, Caldas C, Voest EE. Caring for patients with cancer in the COVID-19 era. Nat Med. 2020 May;26(5):665-671. doi: 10.1038/s41591-020-0874-8. Epub 2020 Apr 16. PMID 32405058
- [Background] Wong ZW, Cross HL. Telehealth in cancer care during the COVID-19 pandemic. Med J Aust. 2020 Sep;213(5):237-237.e1. doi: 10.5694/mja2.50740. Epub 2020 Aug 16. No abstract available. PMID 32803783
- [Background] Dickinson R, Hall S, Sinclair JE, Bond C, Murchie P. Using technology to deliver cancer follow-up: a systematic review. BMC Cancer. 2014 May 3;14:311. doi: 10.1186/1471-2407-14-311. PMID 24885758
- [Background] Finnane A, Dallest K, Janda M, Soyer HP. Teledermatology for the Diagnosis and Management of Skin Cancer: A Systematic Review. JAMA Dermatol. 2017 Mar 1;153(3):319-327. doi: 10.1001/jamadermatol.2016.4361. PMID 27926766
- [Background] Kubendran S, Sivamurthy S, Schaefer GB. A novel approach in pediatric telegenetic services: geneticist, pediatrician and genetic counselor team. Genet Med. 2017 Nov;19(11):1260-1267. doi: 10.1038/gim.2017.45. Epub 2017 Apr 27. PMID 28471436
- [Background] Agha Z, Schapira RM, Laud PW, McNutt G, Roter DL. Patient satisfaction with physician-patient communication during telemedicine. Telemed J E Health. 2009 Nov;15(9):830-9. doi: 10.1089/tmj.2009.0030. PMID 19919189
- [Background] Hennemann-Krause L, Lopes AJ, Araujo JA, Petersen EM, Nunes RA. The assessment of telemedicine to support outpatient palliative care in advanced cancer. Palliat Support Care. 2015 Aug;13(4):1025-30. doi: 10.1017/S147895151400100X. Epub 2014 Aug 27. PMID 25159308
- [Background] Sabesan S, Larkins S, Evans R, Varma S, Andrews A, Beuttner P, Brennan S, Young M. Telemedicine for rural cancer care in North Queensland: bringing cancer care home. Aust J Rural Health. 2012 Oct;20(5):259-64. doi: 10.1111/j.1440-1584.2012.01299.x. PMID 22998200
- [Background] Buchanan AH, Datta SK, Skinner CS, Hollowell GP, Beresford HF, Freeland T, Rogers B, Boling J, Marcom PK, Adams MB. Randomized Trial of Telegenetics vs. In-Person Cancer Genetic Counseling: Cost, Patient Satisfaction and Attendance. J Genet Couns. 2015 Dec;24(6):961-70. doi: 10.1007/s10897-015-9836-6. Epub 2015 Apr 3. PMID 25833335
- [Background] Schwartz MD, Valdimarsdottir HB, Peshkin BN, Mandelblatt J, Nusbaum R, Huang AT, Chang Y, Graves K, Isaacs C, Wood M, McKinnon W, Garber J, McCormick S, Kinney AY, Luta G, Kelleher S, Leventhal KG, Vegella P, Tong A, King L. Randomized noninferiority trial of telephone versus in-person genetic counseling for hereditary breast and ovarian cancer. J Clin Oncol. 2014 Mar 1;32(7):618-26. doi: 10.1200/JCO.2013.51.3226. Epub 2014 Jan 21. PMID 24449235
- [Background] Thaker DA, Monypenny R, Olver I, Sabesan S. Cost savings from a telemedicine model of care in northern Queensland, Australia. Med J Aust. 2013 Sep 16;199(6):414-7. doi: 10.5694/mja12.11781. PMID 24033216
- [Background] Marteau TM, Dormandy E, Michie S. A measure of informed choice. Health Expect. 2001 Jun;4(2):99-108. doi: 10.1046/j.1369-6513.2001.00140.x. PMID 11359540
- [Background] Vadaparampil ST, Quinn GP, Small BJ, McIntyre J, Loi CA, Closser Z, Gwede CK. A pilot study of hereditary breast and ovarian knowledge among a multiethnic group of Hispanic women with a personal or family history of cancer. Genet Test Mol Biomarkers. 2010 Feb;14(1):99-106. doi: 10.1089/gtmb.2009.0088. PMID 19929403
- [Background] Cohn J, Blazey W, Tegay D, Harper B, Koehler S, Laurent B, Chan V, Jung MK, Krishnamachari B. Physician Risk Assessment Knowledge Regarding BRCA Genetics Testing. J Cancer Educ. 2015 Sep;30(3):573-9. doi: 10.1007/s13187-014-0724-9. PMID 25234477
- [Background] Chan V, Blazey W, Tegay D, Harper B, Koehler S, Laurent B, Lipka S, Cohn J, Jung MK, Krishnamachari B. Impact of academic affiliation and training on knowledge of hereditary colorectal cancer. Public Health Genomics. 2014;17(2):76-83. doi: 10.1159/000356938. Epub 2014 Jan 22. PMID 24458016
- [Background] Bannon SA, Mork M, Vilar E, Peterson SK, Lu K, Lynch PM, Rodriguez-Bigas MA, You YN. Patient-reported disease knowledge and educational needs in Lynch syndrome: findings of an interactive multidisciplinary patient conference. Hered Cancer Clin Pract. 2014 Feb 5;12(1):1. doi: 10.1186/1897-4287-12-1. PMID 24499499
- [Background] McAllister M, Wood AM, Dunn G, Shiloh S, Todd C. The Genetic Counseling Outcome Scale: a new patient-reported outcome measure for clinical genetics services. Clin Genet. 2011 May;79(5):413-24. doi: 10.1111/j.1399-0004.2011.01636.x. Epub 2011 Feb 14. PMID 21255005
- [Background] Yuen J, Lee SY, Courtney E, Lim J, Soh H, Li ST, Chen Y, McAllister M, Fenwick EK, Ngeow J. Evaluating empowerment in genetic counseling using patient-reported outcomes. Clin Genet. 2020 Feb;97(2):246-256. doi: 10.1111/cge.13646. Epub 2019 Oct 23. PMID 31571202
- [Background] Grant PE, Pampaka M, Payne K, Clarke A, McAllister M. Developing a short-form of the Genetic Counselling Outcome Scale: The Genomics Outcome Scale. Eur J Med Genet. 2019 May;62(5):324-334. doi: 10.1016/j.ejmg.2018.11.015. Epub 2018 Nov 26. PMID 30496830
- [Background] DeMarco TA, Peshkin BN, Mars BD, Tercyak KP. Patient satisfaction with cancer genetic counseling: a psychometric analysis of the Genetic Counseling Satisfaction Scale. J Genet Couns. 2004 Aug;13(4):293-304. doi: 10.1023/b:jogc.0000035523.96133.bc. PMID 19736695
- [Background] Thomas C, McAllister M. Establishing the minimum clinically important difference for the Genetic Counseling Outcome Scale (GCOS-24). J Genet Couns. 2019 Oct;28(5):1003-1010. doi: 10.1002/jgc4.1152. Epub 2019 Jul 30. PMID 31361378
- [Background] Voils CI, Venne VL, Weidenbacher H, Sperber N, Datta S. Comparison of Telephone and Televideo Modes for Delivery of Genetic Counseling: a Randomized Trial. J Genet Couns. 2018 Apr;27(2):339-348. doi: 10.1007/s10897-017-0189-1. Epub 2017 Dec 15. PMID 29243007
- [Background] Zilliacus EM, Meiser B, Lobb EA, Kelly PJ, Barlow-Stewart K, Kirk JA, Spigelman AD, Warwick LJ, Tucker KM. Are videoconferenced consultations as effective as face-to-face consultations for hereditary breast and ovarian cancer genetic counseling? Genet Med. 2011 Nov;13(11):933-41. doi: 10.1097/GIM.0b013e3182217a19. PMID 21799430